CLINICAL TRIAL: NCT02800018
Title: Evaluation of Perinatal Risk Factors for Hypoxic-ischaemic Encephalopathy (HIE) and Their Influence on Severity of Encephalopathy During and After Hypothermia Therapy
Brief Title: Correlation of Risk Factors and Severity of Hypoxic-ischaemic Encephalopathy
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00242
Record Dates: First submitted 2016-06-03; First posted 2016-06-15 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Hypoxic Ischaemic Encephalopathy
Keywords: hypothermia therapy; perinatal asphyxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: risk factors — investigators will analyze if certain risk factors will influence the progression of the encephalopathy

SUMMARY:
The first aim of this study is to analyse perinatal risk factors leading to hypoxic ischaemic encephalopathy in term and near term neonates born in Switzerland who were admitted to the neonatal and intensive care units offering hypothermia therapy.

Further, investigators would like to analyse the influence of these perinatal risk factors on the severity of encephalopathy during and after hypothermia therapy.

DETAILED DESCRIPTION:
Encephalopathy of the neonate could have different aetiologies. Perinatal asphyxia leading to hypoxia-ischaemia is frequent ,1-2 per 1000 life born neonates are affected. Hypoxic ischaemic encephalopathy is one of the most important causes for adverse neurodevelopmental outcome, cerebral palsy, epilepsy and hearing and vision deficiencies in term and near term neonates. Til now, hypothermia therapy is the only therapy reducing the risk of adverse neurodevelopmental outcome and is nowadays standard of care. In this study investigators would like to analyse perinatal risk factors causing HIE and their influence on the Sarnat Score on day 1 and 3 of life (during hypothermia therapy) and on day 4 of life (after hypothermia therapy).

ELIGIBILITY:
Inclusion Criteria:

* This study includes data of neonates suffering from hypoxic-ischaemic encephalopathy born with a gestational age > 35 0/7 weeks, who were admitted to the neonatal and intensive care units in Switzerland between 2011-2013 and were treated with therapeutic hypothermia.

Exclusion Criteria:

* Neonates with hypoxic-ischaemic encephalopathy, born with a gestational age < 35 0/7 weeks or without hypothermia treatment or syndromal diseases or with malformations were excluded.
* Further, children without consent to research use were excluded.

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates born >35 0/7 gestational weeks with clinical signs of hypoxic encephalopathy with Apgar Score<5 with 10minutes of life, mechanical ventilation with 10minutes of life, pH 7.0 or BE -16mmol/L, lactate >12mmol/L within 60minutes after birth, and seizures or Sarnat staging II-III or Thompson Score >7.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with either antepartal or intrapartal risk factors leading to hypoxic ischaemic encephalopathy and influence of these risk factors on sarnat staging during and after hypothermia therapy | 7 days
  The investigators evaluate the incidence of the known antepartal and intrapartal risk factors and analyze if there is a statistically significant difference of the influence of intrapartal or antepartal risk factors on the progression of the encephalopathy during and after hypothermia therapy. The investigators analyze sarnat staging on day one and three as a subject to the forementioned risk factors.

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scheidegger S, Held U, Grass B, Latal B, Hagmann C, Brotschi B; National Asphyxia and Cooling Register Group. Association of perinatal risk factors with neurological outcome in neonates with hypoxic ischemic encephalopathy. J Matern Fetal Neonatal Med. 2021 Apr;34(7):1020-1027. doi: 10.1080/14767058.2019.1623196. Epub 2019 Jun 4. PMID 31117854